CLINICAL TRIAL: NCT06497621
Title: Effect of Two Impression Techniques on Retention of Maxillary Complete Denture in Pakistani Population: A Double-blinded Crossover Randomized Controlled Trial
Brief Title: Comparing Impression Techniques for Maxillary Complete Denture Retention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Syed Murtaza Raza Kazmi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023-8450-25606
Record Dates: First submitted 2024-05-03; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Denture Retention; Patient Satisfaction
Keywords: Crossover; Complete Denture; Retention; Poly-vinyl siloxane
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single step PVS impression (Experimental): Single-step final impression method for complete denture fabrication using medium body PVS for border molding and wash impression in a single-step (i.e., one insertion of impression tray in mouth).
  Interventions: Procedure: Single step PVS impression
- Conventional two-step PVS impression (Active Comparator): Two-step final impression method for complete denture fabrication, i.e., border molding with heavy-body PVS first, followed by wash impression with light-body PVS.
  Interventions: Procedure: Conventional two-step PVS impression

INTERVENTIONS:
Procedure: Single step PVS impression — Single-step final impression method for complete denture fabrication using medium body PVS for border molding and wash impression in a single-step (i.e., one insertion of impression tray in mouth).
  Arms: Single step PVS impression
Procedure: Conventional two-step PVS impression — Border molding with heavy-body PVS first, followed by wash impression with light-body PVS
  Arms: Conventional two-step PVS impression

SUMMARY:
The primary objective of this protocol is to compare retention in maxillary complete dentures using single-versus two-step Poly-vinyl Siloxane (PVS) impressions in edentulous patients at denture delivery. Secondary objectives include assessing patient satisfaction with impression methods and denture satisfaction after a two-month adaptation and comparing post-delivery adjustment visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderately resorbed maxillary alveolar ridge
* Patients with bimaxillary edentulous arches
* Patients aged between 35 to 85 years willing to participate in the study
* Patients who could be available for follow up visits

Exclusion Criteria:

* Patients with palatal torus or bony exostoses or severe undercuts in the maxillary arch
* Patients with uncontrolled diabetes, osteoporosis, osteomalacia and osteopenia
* Patients with xerostomia
* Patients with mucosa covering the denture bearing area with signs of inflammation, ulceration, or hyperplasia.
* Patients undergoing radiotherapy or chemotherapy or maxillofacial surgery
* Patients suffering from maxillofacial trauma
* Patients with neuromuscular disorders
* Patients with clinical signs and symptoms of temporomandibular joint dysfunction
* Patients with highly resorbed maxillary ridge and/ or flabby ridge
* Patient with hypersensitivity to silicone materials

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Retention of maxillary denture using digital force meter | At the delivery appointment for each denture at an average of 2.5 week from the start of denture fabrication and at 8th week (+/- 3 days)
  Three readings will be taken for each maxillary denture using digital force meter, and an average will be calculated in units for Newton (N) or Kg.m/s2.

SECONDARY OUTCOMES:
Patient satisfaction with impression methods via the Burdens in Dental Impression-Making Questionnaire (BiDIM-Q) | At the delivery appointment for each denture at an average of 2.5 week from the start of denture fabrication and at 8th week (+/- 3 days)
  The questionnaire consists of 12 questions covering various aspects of the impression-making process. Prosthodontists will request patients to score each question from 1 to 100 to gauge their response. A higher score for an aspect of the impression-making procedure will indicate a higher degree of satisfaction.
Denture satisfaction using the Denture Satisfaction (DS) questionnaire. | At 2 months
  The questionnaire comprises 11 questions, answered on a 4-point Likert-type scale to assess the patient's experience with the dentures provided.

OTHER OUTCOMES:
Number of post-insertion visits for denture adjustment | At the end of adjustment period of each denture at an average of 1-month after denture delivery
  The research team will record the post-delivery visits required to adjust dentures fabricated from two different impression methods in the study Pro-forma.

IPD SHARING:
Plan to Share IPD: No